CLINICAL TRIAL: NCT06736496
Title: Comparative Study of Opioid-Free Anesthesia Versus Opioid Anesthesia in Patients Undergoing Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mokhtar Mohamed, resident doctor at Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Free vs Opioid Anesthesia
Record Dates: First submitted 2024-12-12; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Nalbuphine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (Experimental): patients will receive : nalbuphine administered at a dose of 0.2 mg / kg IV bolus dose before induction and intermittent doses of 0.5 mg/kg if MAP and HR greater than 20% of the base line value.
  Interventions: Drug: Nalbuphine
- group 2 (Experimental): patients will receive : Dexmedetomidine infusion at rate of 0.5mcg/kg/h initiated 10 min before induction and ketamine iv bolus dose of 0.35 mg/kg and Lidocaine iv bolus dose of 1mg/kg administrated before skin incision.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Nalbuphine — patients will receive : nalbuphine administered at a dose of 0.2 mg / kg IV bolus dose before induction and intermittent doses of 0.5 mg/kg if MAP and HR greater than 20% of the base line value.
  Arms: group 1
Drug: Dexmedetomidine — patients will receive : Dexmedetomidine infusion at rate of 0.5mcg/kg/h initiated 10 min before induction and ketamine iv bolus dose of 0.35 mg/kg and Lidocaine iv bolus dose of 1mg/kg administrated before skin incision.
  Arms: group 2

SUMMARY:
Laparoscopic cholecystectomy is an effective surgical approach for the treatment of gallbladder disorders such as cholecystitis, gallbladder stones or gallbladder polyps. Although the surgical technique for the treatment of cholecystitis with laparoscope shows some gains compared to open surgery, postoperative complications such as abdominal incision pain, nausea and vomiting, or other complications are still challenging issues.

Thus, there is a need to study and evaluate new non-opioid pain medications after laparoscopic cholecystectomy as part of an opioid reduction strategy.the aim of the study is To compare the effectiveness and safety of opioid-free anesthesia versus opioid-based anesthesia in patients undergoing laparoscopic cholecystectomy, focusing on pain management, postoperative recovery, and incidence of adverse effects.

DETAILED DESCRIPTION:
Anesthesia requires a full spectrum of drugs, from which an anesthetic plan can be applied to achieve the desired level of sedation, analgesia, amnesia, muscle relaxation, and reflex abolition.

Opioid administration as a bolus dose or continuous infusion is commonly used by anesthesiologists in major and day care surgeries. Using of opioids during anesthesia is associated with various opioid-related adverse effects such as respiratory depression, opioid-induced hyperalgesia, nausea and vomiting, urinary retention, paralytic ileus, and the risk of cognitive and sleep dysfunction , This negative side effect profile of opioids may cause delayed recovery and discharge of patients from the post-anesthesia care unit as well as unanticipated hospital readmissions.

The emergence of opioid-free anesthesia was prompted by the adverse effects of opioids and the ongoing opioid epidemic.

Opioid-free anesthesia is a multimodal anesthetic and analgesic without the use of opioid drugs and can play a crucial role in enhanced recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* o Adults aged 18-65 years.

  * Scheduled for elective laparoscopic cholecystectomy.
  * ASA Physical Status I-III.
  * Provided informed consent.

Exclusion Criteria:

* patients with a history of alcohol or drug abuse.

  * Chronic opioid use or dependence.
  * basal heart rate (HR) ≤ 50 beats/min.
  * Allergies to study medications.
  * Severe renal or hepatic impairment.
  * Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
amount of opioid consumption | 24 hours
  Total opioid consumption in the postoperative period.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blaudszun G, Lysakowski C, Elia N, Tramer MR. Effect of perioperative systemic alpha2 agonists on postoperative morphine consumption and pain intensity: systematic review and meta-analysis of randomized controlled trials. Anesthesiology. 2012 Jun;116(6):1312-22. doi: 10.1097/ALN.0b013e31825681cb. PMID 22546966
- [Background] Collard V, Mistraletti G, Taqi A, Asenjo JF, Feldman LS, Fried GM, Carli F. Intraoperative esmolol infusion in the absence of opioids spares postoperative fentanyl in patients undergoing ambulatory laparoscopic cholecystectomy. Anesth Analg. 2007 Nov;105(5):1255-62, table of contents. doi: 10.1213/01.ane.0000282822.07437.02. PMID 17959952
- [Background] Weibel S, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Afshari A, Kranke P. Efficacy and safety of intravenous lidocaine for postoperative analgesia and recovery after surgery: a systematic review with trial sequential analysis. Br J Anaesth. 2016 Jun;116(6):770-83. doi: 10.1093/bja/aew101. PMID 27199310
- [Background] Loftus RW, Yeager MP, Clark JA, Brown JR, Abdu WA, Sengupta DK, Beach ML. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. Anesthesiology. 2010 Sep;113(3):639-46. doi: 10.1097/ALN.0b013e3181e90914. PMID 20693876
- [Background] Dinges HC, Otto S, Stay DK, Baumlein S, Waldmann S, Kranke P, Wulf HF, Eberhart LH. Side Effect Rates of Opioids in Equianalgesic Doses via Intravenous Patient-Controlled Analgesia: A Systematic Review and Network Meta-analysis. Anesth Analg. 2019 Oct;129(4):1153-1162. doi: 10.1213/ANE.0000000000003887. PMID 30418234